CLINICAL TRIAL: NCT01299545
Title: Validation Study of RA-INF-Dx as a Multigene Molecular Test Intended to Aid in the Identification of Patients With Rheumatoid Arthritis Who Are Unlikely to Show an Initial Response to Infliximab and Methotrexate Combination Therapy
Brief Title: Validation Study of RA-INF-Dx, a Multigene Molecular Test Used to Predict Non-Response to INfliximab Therapy
Acronym: PRINT
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties
Sponsor: TcLand Expression S.A. (Industry)
Collaborators: Premier Research (Other); Theradis pharma (Unknown); Medpharmgene, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010-A01046-33
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Anti TNF; Infliximab; Methotrexate; DMARDs; Gene expression biomarkers
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood sampling in Paxgene tubes (DNA, RNA) Whole blood sampling in EDTA tubes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- a single group of patients -200 expected: polyarthrite rhumatoid patients

SUMMARY:
Study Design & Objectives:

Multi-centre, non-interventional, open-label, non-comparative, prospective cohort study with a clinical follow-up between 12 and 14 weeks.

To determine the performances of the RA-INF-Dx blood test intended to aid in the identification of patients with rheumatoid arthritis who are unlikely to show an initial response to infliximab and methotrexate combination therapy evaluated according to EULAR response criteria.

Ancillary study objective:

To constitute a biocollection of samples associated with all clinical and biological data collected at inclusion and at the evaluation visit.

DETAILED DESCRIPTION:
The RA-INF-Dx test is a non invasive in vitro blood test intended to aid in the identification of patients with RA who are unlikely to show an initial response to infliximab and methotrexate combination therapy.

The RA-INF-Dx test is indicated for use in patients:

* 18 years of age or older,
* Eligible for a first line biologic therapy with infliximab. The RA-INF-Dx test is indicated for use by rheumatologists as a biological basis for guiding infliximab treatment prior to its initiation.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Rheumatoid Arthritis

1. Patient with a confirmed Rheumatoid Arthritis according the American College of Rheumatology (ACR) classification criteria.

   Disease Activity
2. Patient with a DAS28 greater than 3.2.

   Treatment
3. Patient eligible for a first line TNFα blocking agent treatment with infliximab according to the "Summary of Product Characteristics",
4. Patient refractory to treatment with at least one classical DMARDs (one of which has to be MTX) prescribed according to the international recommendations, i.e. for at least 12 weeks at the maximal tolerated dose prior to infliximab treatment and with doses which must have been kept stable during the 4 weeks preceding the initiation of the infliximab therapy (patients may be included if they have undergone a wash-out period using cholestyramine or equivalent subsequent to leflunomide treatment),
5. Use of oral steroids (≤ 10mg/day of prednisone or equivalent dose of another molecule) and/or NSAIDs will be permitted; doses must have been kept stable during the 4 weeks preceding the initiation of the infliximab therapy,

   Other criteria
6. Patient (male or female) at 18 years of age or older at inclusion,
7. Negative β-HCG pregnancy test, when appropriate according to the patient's age and contraceptive method,
8. Informed consent signed.

Exclusion Criteria:

1. Patient having received previous courses of other biologic therapy (TNF blocking agents, anti-CD20, anti-CTLA4, IL1 blockers, IL6 blockers and other molecules in development),
2. Patient non eligible to infliximab therapy according to the "Summary of Product Characteristics",
3. Patient with clinically significant, severe and uncontrolled infectious diseases,
4. Patient with symptoms of a significant somatic or psychiatric/mental illness,
5. Patient with other auto-immune diseases (i.e. Inflammatory Bowel Diseases, Systemic Lupus Erythematosus, vasculitis, uncontrolled asthma, etc...),
6. Patient with evidence of cardiac, pulmonary, metabolic, renal, hepatic, gastro-intestinal conditions, which, in the opinion of the investigator, may interfere with the study,
7. Pregnancy,
8. Patient that is participating in a clinical trial or that participated in a previous one within 10 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from RA eligible to a first biologic therapy for whom the treating rheumatologist envisages infliximab therapy will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To determine the performances of the RA-INF-Dx test to aid in the identification of patients with RA who are unlikely to show an initial response to infliximab and methotrexate combination therapy. | Performed at inclusion : blood samples will be taken before the infliximab infusion.
  Statistical relationship between the RA-INF-Dx blood test results and the non-response (evaluated according to EULAR criteria) to infliximab and methotrexate combination therapy will be analyzed.

SECONDARY OUTCOMES:
Non-response to infliximab and methotrexate combination therapy based on American College of Rheumatology (ACR) criteria | at the time of the first response evaluation (between the 12th and the 14th week)
  A statistical analysis will be performed in order to evaluate the predictive performances of the test validated in the study primary objective in relation to the non-response to infliximab and methotrexate combination therapy evaluated according to ACR criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sara MARSAL, MD, Principal Investigator — University Hospital Val d'Hebron (Barcelona, Spain)
Locations (37):
- Canada (5):
  - Location n°31, Mississauga - Chow
  - Location n°36, Ontario
  - Location n°34, Rimouski
  - Location n°33, Saskatchewan
  - Location n°35, Toronto
- France (8):
  - Location n°41, Amiens
  - Location n°13, Bobigny
  - Location n°39, Dreux
  - Location n°14, Grenoble
  - Location n°40, Meaux
  - Location n°25, Paris
  - Location n°37, Paris (Hop Bichat)
  - Location n°38, Strasbourg
- Hungary (5):
  - Location n°6, Budapest
  - Location n°8, Budapest
  - Location n°7, Debrecen
  - Location n°10, Eger
  - Location n°9, Kistarcsa
- Italy (3):
  - Location n°15, Messina
  - Location n°16, Milan
  - Location n°17, Pisa
- Lithuania (4):
  - Location n°27, Kaunas
  - Location n°29, Klaipėda
  - Location n°30, Panevezys
  - Location n°28, Vilnius
- Romania (8):
  - Location n° 19, Bucharest
  - Location n°20, Bucharest
  - Location n°22, Bucharest
  - Location n°23, Bucharest
  - Location n°21, Cluj-Napoca
  - Location n°24, Iași
  - Location n°26, Iași
  - Location n°18, Timișoara
- Slovakia (2):
  - Location n°12, Banská Bystrica
  - Location n°11, Piešťany
- Spain (2):
  - Location n°3, Málaga
  - Location n°5, Oviedo